CLINICAL TRIAL: NCT00083525
Title: Urokinase-Plasminogen Activator (uPA) Inhibitor WX-UK1 in Combination With Capecitabine in Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Heidelberg Pharma AG (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WX/50-005
Record Dates: First submitted 2004-05-25; First posted 2004-05-26 (Estimated); Last update posted 2008-01-24 (Estimated); Status verified 2008-01

CONDITIONS: Advanced Malignancies
MeSH Terms: interventions — N-alpha-(2,4,6-triisopropyl-phenylsulfonyl)-3-amidino-(L)-phenyl-alanine-4-ethoxycarbonyl-piperazide hydrochloride; Capecitabine

INTERVENTIONS:
Drug: WX-UK1 in combination with Capecitabine

SUMMARY:
The purpose of this study is to determine the safety, tolerability, maximum tolerated dose (MTD), pharmacokinetics, and pharmacodynamics of the combination of WX-UK1 and capecitabine in patients with advanced malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of a non-hematologic malignancy that is either unresponsive to currently available therapies or for which there is no known effective therapy.
* Patient willing to give informed consent, understand and comply with study procedures/restrictions
* Age>=18
* Patients must have an ECOG performance status of 0, 1, or 2
* Life expectancy of > 12 weeks
* Negative serum pregnancy test for women of child-bearing potential and not nursing. Fertile patients must use effective contraception during and for 30 days (women) or 4 months (men) after treatment with WX-UK1.
* Measurable or non-measurable disease. Patients without clinical or radiologic evidence of disease are not eligible.
* Laboratory parameters (obtained within the screening period): WBC >= 3 G/L, neutrophils >= 1.5 G/L, platelets >= 100 G/L, Hgb >= 9 g/dL), total bilirubin <= 1.5 x ULN, ASAT/ALAT/AP/GGT <= 2.5 x ULN, serum creatinine <= 2 x ULN.

Exclusion Criteria:

* History of hypersensitivity to the study drugs or chemically related compounds or any of the excipients
* History of or current neurological disorder, in particular an active or treated seizure disorder
* Known standard therapy for the patient's disease that is potentially curative or known to extend life expectancy.
* Carcinomatous meningitis or untreated/uncontrolled metastatic brain parenchymal disease.
* Concurrent or prior (within 4 weeks prior to start of WX-UK1 treatment for cytotoxic chemotherapy, biological-, endocrine-, investigational- or radiotherapy and 6 weeks for nitrosoureas, mitomycin-C)
* Uncontrolled infection
* Significant cardiac disease (NYHA classification III or IV
* Contraindication to an infusion volume of 1000 ml over 2 h
* History of or current blood coagulation disorders
* History of or current bleeding disorder (including cerebral bleeding, recurrent massive nose bleeds, hematuria or unexplained bruising)
* Diabetes mellitus, if not controlled by insulin, oral anti-diabetic agents or diet alone
* Anticoagulant or thrombolytic therapy within four weeks prior to start of treatment (except heparin flush to keep a port open or coumadin 1 mg/day or ASA 100mg/d)
* Active serious illness that renders the patient unsuitable for study entry or multiple blood sampling
* Illness or condition that might alter the absorption, distribution, metabolism and elimination of WX-UK1
* Known Hepatitis B/C or HIV infection
* Contraindication to capecitabine intake as specified in the SPC such as DPD-deficiency or concomitant intake of sorivudine or sorivudine related compounds
* Known hemorrhagic brain metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2004-05

CONTACTS AND LOCATIONS:
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States